CLINICAL TRIAL: NCT04696796
Title: Comparison of Episiotomy Scissors and BasIQ-4 Episiotomy Device in Mediolateral Episiotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-9.1/45
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Episiotomy Wound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BasIQ-4 Surgical Knife (Experimental): Following the administration of 10 ml of 1% lidocaine, mediolateral episiotomy will be preformed with BasIQ-4 Surgical Knife according to computer generated randomization.
  Interventions: Procedure: Mediolateral Episiotomy with BasIQ-4 Surgical Knife
- Episiotomy Scissors (Active Comparator): Following the administration of 10 ml of 1% lidocaine, mediolateral episiotomy will be preformed with episiotomy scissors according to computer generated randomization.
  Interventions: Procedure: Mediolateral Episiotomy with Episiotomy Scissors

INTERVENTIONS:
Procedure: Mediolateral Episiotomy with BasIQ-4 Surgical Knife — Mediolateral episiotomy will be performed with BasIQ-4 Surgical Knife which cuts from distal to the center with inner knife.
  Arms: BasIQ-4 Surgical Knife
Procedure: Mediolateral Episiotomy with Episiotomy Scissors — Mediolateral episiotomy will be made from the central to the distal with episiotomy scissors
  Arms: Episiotomy Scissors

SUMMARY:
Episiotomy is an obstetric intervention performed to facilitate, accelerate and / or prevent third and fourth degree perineal tears by cutting the vagina at the end of the second stage of labor. Postpartum perineal pain affects patients' lives significantly and causes negative effects on work life, social life and family relations. Median episiotomy is associated with 3-4 times increased anal sphincter injury as well as easy recovery. Therefore, mediolateral episiotomy is preferred in Europe. The common feature was that scissors are used in previous studies and the incision was made from the central to the distal. A randomized controlled clinical study is planned to compare the scissors and episiotomy device BasIQ-4, which carries scalpel, holding apparatus, and cuts from distal to the center in mediolateral episiotomy. This is the first study in humans in this field.

DETAILED DESCRIPTION:
Pregnant women who applied to Ege University Gynecology and Obstetrics Department Delivery Room Service and had vaginal delivery will be included in the study after obtaining their consent. When the cases meeting the inclusion criteria will be taken to the delivery table for delivery, verbal consent will be obtained by the physician if the need for episiotomy is determined by the physician in the second stage of delivery. Following the administration of 10 ml of 1% lidocaine, mediolateral episiotomy will be opened with scissors or Basiq-4 according to computer generated randomization. The presence of shoulder dystocia during delivery, the number of moves for episiotomy incision, the duration of stage 2, fetal weight, the degree of perineal injury, any additional injury, and urethral injury will be recorded in the prepared case form. Then, the episiotomy incision will be continuously sutured with 2-0 slow dissolving polyglactin 910 suture material for all cases.

The length of episiotomy after suturing and the length of perineal injury, if any, will be measured with a sterile ruler and recorded on the case form. Postpartum discharge is carried out 48 hours after birth in accordance with the Ministry of Health Regulations. Participants will be reassessed during discharge in terms of pain with the Visual Pain Scale (VAS).

The cases will be evaluated by the study team again, and notes regarding episiotomy length, infection, pain, incision separation, fecal incontinence, rectovaginal fistula, and painful defecation will be recorded on the case form six months after delivery. Participants will be requested to fill FSFI forms to evaluate their sexual lives.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous singleton pregnancies > 37th gestational week
2. Estimated fetal weight between 3000-4000g
3. The need for an episiotomy in the second stage of labor
4. Vertex presentation

Exclusion Criteria:

1. Additional internal disease
2. Inability to communicate in Turkish and English
3. Multiple pregnancy
4. Episiotomies in emergency situations without crowning the baby's head
5. Using vacuum device at birth

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Pain Assessed by VAS at 48 Hours After Birth | 48 hours
  Participants will be reassessed during discharge in terms of pain with the Visual Pain Scale (VAS). The participants will asked to rate current pain on a 10-cm visual analog scale (VAS), with 0 being no pain and 10 the worst pain imaginable 48 hours after operation.
FSFI Score | 6 months
  Participants will be requested to fill FSFI (Female Sexual Function Index) forms to evaluate their sexual lives six months after birth. The FSFI consists of 19 questions and is a validated questionnaire for the assessment of sexual function. The questions are grouped into the domains of libido, arousal, lubrication, orgasm, satisfaction, and pain. Higher scores reflect better sexual function (maximum score 36), including pain, in which 0 reflects lots of pain and 5 reflects the absence of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Hospital, Izmir, Bornova, Turkey (Türkiye)